CLINICAL TRIAL: NCT01660620
Title: Topical Betaxolol for the Prevention of Retinopathy of Prematurity
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Smith-Kettlewell Eye Research Institute (Other)
Collaborators: Ohio State University (Other); University of Minnesota (Other); University of Oklahoma (Other); The University of Texas Health Science Center, Houston (Other)
Responsible Party: Principal Investigator, William V Good, MD, Administrator, Smith-Kettlewell Eye Research Institute
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 108298
Record Dates: First submitted 2012-08-06; First posted 2012-08-08 (Estimated); Last update posted 2013-01-03 (Estimated); Status verified 2012-08

CONDITIONS: Development of Side Effects From Betaxolol
Keywords: betaxolol/ retinopathy of prematurity
MeSH Terms: interventions — Betaxolol

STUDY DESIGN:
Who Masked: Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- betaxolol (Experimental): betaxolol 0.25% 2 per day for 3 weeks
  Interventions: Drug: Betaxolol
- placebo (Placebo Comparator): masked labeling also 2 per day administration
  Interventions: Drug: topical betaxolol

INTERVENTIONS:
Drug: Betaxolol
  Arms: betaxolol
Drug: topical betaxolol — given topically
  Arms: placebo

SUMMARY:
We hypothesize that topical betaxolol will reduce the development of severe retinopathy of prematurity.

DETAILED DESCRIPTION:
The drug is administered twice a day between 32 and 35 weeks gestational age, at a t ime when ROP is most likely to arise.

ELIGIBILITY:
Inclusion Criteria:

* <1251 grms birth weight

Exclusion Criteria:

* ocular defect

Ages: 32 Weeks to 32 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 23 (Actual)
Dates: Start 2011-04; Primary Completion 2011-11 (Actual); Study Completion 2011-11 (Actual)

PRIMARY OUTCOMES:
development of apnea and or bradycardia | 3 weeks
  babies were monitored and HR/RR monitored and recorded by masked observers, periodically

SECONDARY OUTCOMES:
development of ROP requiring treatment | 7 weeks
  Type I ROP was used as a secondary outcome measure